CLINICAL TRIAL: NCT05839366
Title: Adjunctive Esketamine for Analgesia in Mechanically Ventilated ICU Septic Shock Patients
Brief Title: Adjunctive Esketamine for Analgesia in Mechanically Ventilated Septic Shock Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NFEC-2022-394
Record Dates: First submitted 2023-03-20; First posted 2023-05-03 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Septic Shock; Mechanical Ventilation Complication
Keywords: Esketamine; Vasoactive drugs; sedation; analgesia
MeSH Terms: conditions — Shock, Septic; Agnosia | interventions — Esketamine; Sodium Chloride; Saline Solution; Remifentanil; Propofol

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remifentanil + propofol + esketamine (Active Comparator): esketamine (2ml; 50mg), Remifentanil Hydrochloride for Injection (1mg;), propofol injection (50ml; 0.5g; )； The frequency of use is determined by responsible clinicians.All analgesic and sedative drugs used are adjusted according to the actual situation of the patient.
  Interventions: Drug: Esketamine; Drug: Remifentanil + propofol; Procedure: Pain and Sedation Assessment
- remifentanil + propofol + saline (Placebo Comparator): Remifentanil Hydrochloride for Injection (1mg;), propofol injection (50ml; 0.5g; )； The amount of saline used is equivalent to the amount of esketamine.All analgesic and sedative drugs used are adjusted according to the actual situation of the
  Interventions: Drug: Saline; Drug: Remifentanil + propofol; Procedure: Pain and Sedation Assessment

INTERVENTIONS:
Drug: Esketamine — Load dose of 0.25 mg/kg, and the fixed infusion rate of 0.15 mg/kg/h.The load dose will be injected intravenously within 1-2 minutes.Maintain the infusion at a fixed rate of 0.15 mg/kg/h for 72 hours; after 72 hours, change to a fixed rate infusion of 0.06 mg/kg/h.
  Preparation: 46ml of saline + 4ml of eskeamine.
  Other Names: Esketamine Hydrochloride Injection
  Arms: Remifentanil + propofol + esketamine
Drug: Saline — As a placebo,normal saline at the same dose as esketamine.Saline is also administered intravenously.
  Other Names: physiological saline; saline solution
  Arms: remifentanil + propofol + saline
Drug: Remifentanil + propofol — Remifentanil + propofol
Procedure: Pain and Sedation Assessment — RASS Score:
  After randomization success, a baseline Richmond Agitation-Sedation Scale (RASS) score is obtained before administering the investigational drug. Pain assessments are conducted every 1 hour within the first 6 hours after the initiation of the intravenous loading dose of the investigational drug, every 4 hours within the first 24 hours, and subsequently every 8 hours until the end of the study. In addition to the fixed time points mentioned above, researchers may conduct RASS scoring at any time based on the subject's actual condition (excessive or inadequate sedation). (No further RASS scoring is performed once the subject is fully awake.)
  CPOT Score:
  CPOT（Critical-Care Pain Observation Tool）Pain assessments are conducted concurrently with RASS scoring.

SUMMARY:
Sedation and analgesia in patients with sepsis and hemodynamic instability may be challenging in the ICU. Opioids and propofol can further exacerbate tissue infusion in septic shock by reducing cardiac contractility, increasing vasodilation, and reducing respiratory drive. Ketamine is an NMDA receptor antagonist, which has no effect on respiratory drive and has diastolic airway smooth muscle and anti-inflammatory properties. Esketamine is a dextrorotatory cleavage twice as potent and reduces the incidence of dose-dependent side effects of ketamine. Although it has been successfully used in burn patients undergoing multiple operations and anesthesia-related maintenance analgesia, it has not been reported in ICU septic shock patients undergoing mechanical ventilation. The purpose of this study was to explore the use of esketamine in mechanically ventilated ICU septic shock patients in a single-center randomized controlled trial.

DETAILED DESCRIPTION:
In order to further clarify whether Esketamine can be used as a conventional continuous intravenous infusion drug in the ICU, further RCT is required. Therefore, this project assumes that low-dose Esketamine has a clear analgesic and sedative effect, and has advantages such as less adverse reactions in hemodynamics, respiratory inhibition, and gastrointestinal peristalsis. It is proposed to complete the following work: on the standard analgesia and sedation scheme (remifentanil+propofol), evaluate the feasibility, effectiveness and safety of the auxiliary analgesia scheme added with esketamine for septic shock patients with mechanical ventilation by whether to load small dose of esketamine for infusion, so as to provide basis for follow-up individualized diagnosis and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18;
* A patient diagnosed with septic shock;
* It needs to be treated with analgesics, sedatives, and vasopressors for a period of not less than 48 hours;
* Mechanical ventilation by the ventilator is needed;
* Obtain the informed consent of the human subjects or their legal representatives;

Exclusion Criteria:

* Currently pregnant or breastfeeding;
* Confirmed acute severe intracranial or spinal neurologic diseases caused by vascular, intracranial expansion, or injury;
* History of uncontrolled or malignant hypertension (sustained (>3 hours) heart rate >150 beats/min or systolic blood pressure >180 mmHg); recent history of ketamine use；
* Hearing or vision loss, or any other conditions likely to severely interfere with the collection of research data;
* Long-term use of benzodiazepines or opioids;
* Known allergy to any investigational drug;
* Subject receiving sedative therapy not for tolerance to mechanical ventilation (e.g., seizures);
* Unlikely to require ongoing sedation during mechanical ventilation (e.g., Guillain-Barré syndrome);
* Patients deemed unlikely by the attending physician to be weaned from mechanical ventilation, such as those with diseases/injuries primarily affecting respiratory neuromuscular function and conditions requiring prolonged ventilatory support, which are clearly irreversible (e.g., high spinal cord injury);
* Open eye injury or other ophthalmic diseases;
* Concurrent participation in any other interventional study (any study assigning subjects to different treatment groups and/or conducting unconventional diagnostic or monitoring procedures).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2023-05-31 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Doses of remifentanil and norepinephrine during mechanical ventilation (total dose/duration of use hours). | During mechanical ventilation procedure (From randomization to the seventh day of infusion or ventilator withdrawal, whichever occurs first）
  Responsible researchers consult the patient's medical record after completing treatment to obtain the dosage and duration of medication.

SECONDARY OUTCOMES:
Duration of mechanical ventilation. | From endotracheal intubation to withdrawal from mechanical ventilation, or until 28 days after discharge, death, or randomization in the ICU, whichever occurs
  Responsible researchers obtain information by viewing electronic medical records.
Mechanical ventilator free days. | Days to 28
  Responsible researchers obtain information by viewing electronic medical records.
Propofol dosage (total dose/duration of use) during mechanical ventilation. | During mechanical ventilation procedure (From randomization to the seventh day of infusion or ventilator withdrawal, whichever occurs first）
  Responsible researchers consult the patient's medical record after completing treatment to obtain the dosage and duration of medication.
The proportion of patients meeting the RASS sedation and CPOT pain goals during mechanical ventilation. | up to 28 days
  Professionally trained researchers perform RASS and COPT scores on patients at specific time points.
The incidence of delirium, i.e. the positive rate of CAM-ICU. | up to 28 days
  The occurrence of delirium in patients will be recorded by clinicians or nurses on medical records, and researchers will summarize the occurrence of delirium (such as the time of occurrence, duration, treatment measures, etc.)Patients will be evaluated using CAM-ICU by clinicians or nurses.
Incidence of adverse events. | up to 28 days
  The occurrence of adverse events during the hospital period will be recorded in the medical record by the clinician or nurse, and the researcher will obtain the occurrence of adverse events (event type, time, treatment, results, etc.) through the medical record.
Length of ICU stay. | up to 28 days
  Researchers obtain it through the hospital electronic system.
The mortality rate | up to 28 days
  Researchers obtain it through the hospital electronic system.

CONTACTS AND LOCATIONS:
Locations (1):
- Southern medical university Nanfang hospital, Guangzhou, China

IPD SHARING:
Plan to Share IPD: Undecided